CLINICAL TRIAL: NCT04791371
Title: Role of Microvascular Insulin Resistance and Cardiorespiratory Fitness Diabetes
Acronym: REACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Virginia (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-2723; R01DK124344 (NIH)
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; Overweight and Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 Diabetes (Experimental): Participants aged 30-55 with type 2 diabetes
  Interventions: Behavioral: Cardiovascular exercise
- Healthy overweight control (Experimental): Participants aged 30-55 with BMI 25-40 without type 2 diabetes
  Interventions: Behavioral: Cardiovascular exercise

INTERVENTIONS:
Behavioral: Cardiovascular exercise — 15 weeks of cardiovascular exercise 3x/week for 50 minutes/session

SUMMARY:
The goal of this two-site grant proposal is to determine the role of the decreased insulin-mediated muscle perfusion found in type 2 diabetes in contributing to the development of cardiac and skeletal muscle dysfunction and subsequent functional exercise impairment. In addition, it is also our goal to determine whether exercise training attenuates insulin resistance and restores insulin-mediated perfusion to the heart and to skeletal muscle, leading to improved cardiac function and exercise performance.

DETAILED DESCRIPTION:
It is our goal to determine whether exercise training attenuates insulin resistance and restores insulin-mediated perfusion to the heart and to skeletal muscle, leading to improved cardiac function and exercise performance. Data from our two research teams suggest that the cardiac and skeletal muscle microvascular dysfunction present in people with type 2 diabetes contributes to limitations in cardiac and skeletal muscle function associated with impaired functional exercise capacity (a major predictor of CV and all-cause mortality). Insulin action is a potent predictor of the functional exercise capacity impairment in type 2 diabetes. The exact relationship between insulin action, cardiac and muscle dysfunction, cardiac and skeletal muscle perfusion and decreased functional exercise capacity in type 2 diabetes remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (defined as less than 1 hour per week of physical activity)
* BMI: 25-40
* Men and women with and without type 2 diabetes

Exclusion Criteria:

* Documented cardiovascular disease
* Uncontrolled hypertension: disease systolic blood pressure (SBP) > 150, diastolic blood pressure (DBP)> 110
* Obstructive pulmonary disease or asthma
* Peripheral neuropathy
* Physical impairment that would limit exercise ability
* Subjects taking beta blockers, calcium channel blockers, insulin, or Thiazolidinediones (TZD)
* Current or past smoking within the last 1 years
* Current tobacco use
* Anemia
* Control HbA1c > 5.7, T2DM HbA1c > 9
* Pregnant, nursing or hormonal therapy (other than contraceptives)
* Peri or post-menopausal women
* Type 1 diabetes
* Hepatic or renal disease.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in peak oxygen consumption (VO2) | Through study completion, approximately 4 months
  Subjects' peak oxygen consumption will be tested on a stationary bike before and after 15 weeks of exercise
Change in insulin sensitivity | Through study completion, approximately 4 months
  The investigators will evaluate the changes in insulin sensitivity utilizing a euglycemic insulin clamp

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado, Aurora, Colorado
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Park S, Englund EK, Fujiwara T, Enge D, Schafer M, Gerstner Saucedo J, Clark EW, Abushamat LA, Scalzo RL, Fonseca B, Hunter KS, Sammel MD, Regensteiner JG, Reusch JEB, Barker AJ. Comprehensive CMR evaluation including 4D flow-derived E/A vorticity ratio in overweight adults with and without type 2 diabetes mellitus. Cardiovasc Diabetol. 2025 Dec 8;25(1):7. doi: 10.1186/s12933-025-02999-9. PMID 41361416